CLINICAL TRIAL: NCT02909894
Title: Investigating Whether Breaking up Sedentary Behaviour With Seated Upper Body Contractile Activity Can Regulate an Individual's Metabolic Health.
Brief Title: Arming Health: Can Breaking up Restful Sitting Time With Upper Body Contractile Activity Regulate Metabolic Health.
Acronym: AYH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leicester (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0548
Record Dates: First submitted 2016-09-02; First posted 2016-09-21 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2016-08

CONDITIONS: Diabetes
Keywords: Sedentary behaviour; Postprandial glycaemic response
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prolonged Sitting (Experimental)
  Interventions: Other: Prolonged Sitting
- Light intensity arm ergometry breaks (Active Comparator)
  Interventions: Other: Light arm ergometry breaks

INTERVENTIONS:
Other: Prolonged Sitting — Condition A is referred to as the 'sitting' condition. Here participants will remain seated throughout the whole of the 7 ½ hour test period (8am - 3:30pm). On arrival, participants will have a cannula (a small tube that allows us to take blood) inserted into their arm; this will stay in the arm and allow investigators to take regular blood samples throughout the day. Blood samples and blood pressure will be taken at 30, 60, 120 and 180 minutes after breakfast. Following this, a lunch meal will be provided and investigators will continue taking blood samples and blood pressure at 30, 60, 120 and 180 minutes after this lunch meal. In total, 10 blood samples will be taken over the 7 ½ hour testing period. There will also be a cognitive test in the morning and afternoon.
  Arms: Prolonged Sitting
Other: Light arm ergometry breaks — Condition B is the 'light activity breaks' condition. Participants will go through exactly the same process as condition A but will also be asked to do 5 minute bouts of light intensity arm ergometry on a desktop arm ergometer every 30 minutes following breakfast and lunch. In total they will do 12 five minute arm ergometry breaks throughout the 7 ½ hour test period (60 minutes of arm ergometry in total). In total 10 blood samples will be taken on the day.
  Arms: Light intensity arm ergometry breaks

SUMMARY:
Research shows that sitting for long periods of time on a regular basis is bad for health and can leave individuals more susceptible to Obesity, Cardiovascular Disease, Type 2 Diabetes and premature death regardless of exercise engagement outside of these seated hours.

As sitting is so common in modern society it is vital that research explores ways to protect individuals from this worsening issue. Investigators want to see if breaking up long periods of sitting time with short, frequent bouts of light physical activity, while remaining seated, is enough to alleviate these risk factors.

DETAILED DESCRIPTION:
- Familiarisation screening visit - (Visit 1) Before participating in the study, all participants will visit the exercise laboratory for a familiarisation and screening visit where they will be shown the designated experimental area, provide written informed consent and have various measurements taken.

All participants will be required to fast from 10pm onwards the evening prior to this first visit (drinking water is allowed). Participants will then be provided with a standardised breakfast on arrival (after consent has been obtained). This meal will be prescribed according to body mass and will provide approximately 8 kcals per kg of bodyweight made up of 13-14% protein, 51-52% carbohydrate and 35% fat. Typical ingredients used here will be; Plain bagels with margarine and a protein powder mixed with whole milk.

Alternative ingredients matching the nutritional content of this meal will be explored in light of special dietary preferences (i.e. vegan) or food allergies (i.e. lactose intolerance).

It is also important that participants avoid general exercise and drinking alcohol or coffee in the 48 hours (2 days) leading up to this first visit (and the remaining two visits), this will be made clear in the participant information sheet. Very strenuous exercise must be avoided 72 hours (3 days) prior.

Participants will be asked to record all food and drink consumed the day before this first visit. They will then be asked to replicate this diet the day before the remaining visits using their dietary record to guide them. Therefore, all meals leading up to each visit will be standardised and will not confound the results.

The measurements taken during this visit include; basic anthropometry (body mass, waist circumference, body fat %); blood pressure; biochemical variables (HbA1c and blood lipids and CRP); Energy expenditure (at rest, during slow steady state treadmill walking and at numerous intensities on an arm ergometer machine); and measures of objectively determined free-living physical activity, sedentary behaviour and posture.

Anthropometry measurement at visit 1 Arterial blood pressure will be measured in the sitting position. Three measurements will be obtained and the average of the last two measurements will be used.

Basic anthropometric measures such as body mass and body fat percentage (measured through bio impedance analysis) will be taken alongside height and waist circumference (midpoint between the lower costal margin and iliac crest). These will be recorded to the nearest 0.1kg, 0.5%, 0.5cm and 0.5cm respectively.

Biochemical variables collected at visit 1 During visit one a blood sample will be taken whereby HbA1c (Glycated Haemoglobin), CRP (C-Reactive Protein) and lipid profile will be measured. All venepuncture will be undertaken by trained health care professionals and all biochemical analyses will be conducted blinded to treatment condition. All participants will be sent an individual results letter highlighting their main clinical results after the familiarisation visit. With the participants consent, all results will be copied to their GP. Any participant whose Hba1c is 6.5% or above will be sent an individual results letter strongly advising them to make an appointment with their GP as soon as possible to discuss their results in more detail, as this is indicative of Diabetes. Similarly, any participant whose HbA1c is between 6 and 6.4% will also be sent an individual results letter advising them to make an appointment with their GP if they are concerned, as this is indicative of pre-diabetes. With the participants consent, the GP will also be notified of the situation and sent a results letter

Energy Expenditure testing during visit 1 During visit one, the energy expenditure at rest, while walking at 3km/hr and while performing arm ergometry at different intensities will be measured via respiratory gas collected from the participants using the Cortex or GEM breath-by-breath automated gas-analysis system.

In order to assess resting energy expenditure, each participant will be asked to sit quietly (refraining from movement) for 30 minutes while wearing a gas mask/hood. Expired gas data will then be collected over the latter half of this 30 minute period once values have stabilised.

Following this, walking will be performed at 3km.hr on a treadmill for 10 minutes (also while wearing a gas mask), from which expired gas data will be collected in the latter 5 minutes.

Light arm ergometry while seated will then be performed at 5 minute intervals (across numerous intensities) from which expired gas data will be collected in the 2nd 3rd and 4th minutes, discarding both the first and last minute. Participants will also remove the face-mask for 5minutes in between each 5 minute bout in order to allow participants to recover and for energy expenditure outputs to return to their resting level prior to the next activity bout.

This data will consequently dictate the intensity of arm ergometry to be performed when breaking up sitting time, as investigators would like the energy expenditure of these seated breaks to closely resemble that of light walking. This allows investigators to further elucidate the role of posture alone as energy expenditures will be kept relatively consistent with that of previous research, allowing direct comparisons to be made.

Objective measures of physical activity at visit 1 Participants will be issued with an Actigraph accelerometer to measure the time spent sedentary and in moderate to vigorous physical activity under free-living conditions. Participants will be asked to wear this accelerometer (placed on right anterior axillary line) for 7 days after the familiarisation visit, up to 7 days leading up to the treatment conditions and throughout the experimental conditions in order to monitor any potential changes in physical activity levels and make sure participants have avoided exercise in the days leading up to the treatment conditions. Outputs will include steps per day, total body movement (counts per day), and time in sedentary, light, moderate and vigorous-intensity physical activity as determined by counts per minute cut points proposed by Freedson et al. (21)

Posture and sedentary time data collection at visit 1 Postural allocation (sitting and standing) and walking will be quantified using an activPAL physical activity monitor (PAL Technologies, Glasgow, Scotland). The activPAL is a single-unit monitor based on a triaxial accelerometer that is worn midline on the anterior aspect of the thigh and attached directly onto the skin using medical dressing. The monitor produces a signal related to thigh inclination and has been shown to be a valid and reliable measurement tool for determining posture during activities of daily living in a healthy population (22). Outputs from this device include; time spent sitting, standing, stepping and sit-to-stand transitions. The device will be worn for 7 days after the familiarisation visit, (alongside the Actigraph) and throughout experimental conditions.

- Experimental treatment conditions (Visits 2 and 3) In the weeks following this initial familiarization visit, participants will be assigned to receive the following two treatment conditions (A: Prolonged sitting and B: Light arm ergometry breaks) in a random order using an online randomisation tool. Each treatment condition will be carried out on one single day. In total, the study requires three separate visits to the Leicester Diabetes Centre, Leicester General Hospital, University Hospitals of Leicester; familiarisation visit, first treatment condition and second treatment condition.

Where participants have limited access to motorised transport, taxis will be provided to reduce ambulatory activity involved in the commute to and from each visit.

For male participants, there will be a minimum of 7 days between each treatment condition. For females, there will be a gap of one month (or near as possible) due to the potential that different phases of a women's menstrual cycle may affect their blood glucose response to a meal (23). Testing at similar times of the month avoids this potential variability. However, if a female participant reports being post-menopausal on their pre-screening questionnaire then a minimum of 7 days between treatment conditions will be used.

Treatment Condition A: Prolonged sitting During the prolonged sitting condition, participants will be restricted from walking and standing. They will be in a designated room equipped with a chair/desk and have access to a computer with internet services, books and magazines or movies throughout the day. Lavatory breaks will be permitted and a wheelchair will be used to wheel the participants to the toilet to reduce upright activity.

The day before each treatment condition, participants will be asked to consume the same type and quantity of food and drink that they recorded prior to their familiarisation visit. Participants will also be asked to avoid alcohol, caffeine and moderate intensity exercise for 2 days prior to each treatment condition (as done prior to visit one) as reproducibility data has shown that insulin and triglyceride responses to meal ingestion are good under these conditions (24). Furthermore, there is evidence that the effect of a single exercise session on insulin sensitivity and glucose tolerance may last up to 48 hours (25). Strenuous exercise should be avoided for 3 days prior to each treatment condition, as this has been found to increase insulin sensitivity for up to 72 hours (26).

Participants will be asked to fast the night before both treatment conditions (and prior to familiarisation as discussed previously) from 10pm onwards. On the morning of the test, participants will have a cannula inserted into an accessible vein by a trained health care professional and the first of the blood samples will be taken (this represents time point: -1hr according to figure 1). Blood pressure measurements will be taken immediately before each blood sample alongside self-reported measures of positive affect, mood and sleepiness (see description under secondary outcomes section 3.0). Once the cannula has been inserted and the first blood sample taken, participants will then be asked to sit quietly for 60 minutes in order to achieve a steady state. During this time, participants will be expected to complete a battery of cognitive function tests lasting approximately 25 minutes (see description under secondary outcomes section 4.0).

Following this 60 minute period, participants will have another blood pressure measurement, positive affect, mood and sleepiness assessment and blood sample taken, at which point they will then be provided with a standardised mixed meal breakfast (09:00am) (time point: 0h). The meal will be prescribed according to body mass and will provide approximately 8kcals per kg of bodyweight made up of 13-14% protein, 51-52% carbohydrate and 35% fat. A mixed-meal of this nature will be used to ensure ecological validity as fat and carbohydrates are usually co-ingested in real-life situations. Blood sampling alongside positive affect, mood, sleepiness and blood pressure measurements will continue at 30, 60, 120 and 180 minutes following breakfast. A second, lunch meal (12:00pm) (with identical nutrient composition to breakfast), will then be consumed over 15 minutes. Blood pressure, positive affect, mood, sleepiness and blood sampling will continue at 30, 60, 120 and 180 minutes following lunch (Figure 1). Participants will then repeat the battery of cognitive function tests after their final blood sample is taken. All participants will remain sitting throughout the test period whilst undertaking typical sedentary pursuits such as watching TV/DVDs/reading.

Treatment Condition B: Light arm ergometry breaks This will be identical to the prolonged sitting condition (Treatment A), but participants will be required to break up their restful sitting time with seated upper body contractile activity. This will be implemented in the form of arm ergometry breaks for 5 minutes every 30 minutes following both breakfast and lunch. In total, individuals will accumulate 12 bouts (60 minutes) of light intensity arm ergometry.

The main reason for utilising 5 minute bouts every 30 minutes was to achieve a balance between frequency and utility, as having to interrupt sitting time too regularly has less real world application, especially in an office based environment where prolonged sitting is most prevalent. Previous research has also found positive findings while interrupting sitting time in this manner (38).

The intensity (speed and resistance) of these arm ergometry breaks will have been derived from the energy expenditure tests conducted in visit 1, as investigators are aiming to match the intensity of arm ergometry to that of light walking at 3km/hr.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Body Mass Index: ≥ 30 kg/m2
* Male and Female
* Aged: ≥ 30 to ≤ 75 years of age.
* Inactive (I.e. no habitual structured exercise).
* Participant is able to walk (without any assistive devices)

Exclusion Criteria:

* • Aged < 30 or > 75 years of age.

  * Physical condition which limits full participation in the familiarisation visit or treatment visits.
  * Active psychotic illness or other significant illness which, in the view of the investigators, would prevent full participation
  * Inability to communicate in spoken English
  * Steroid use
  * Known Type 2 Diabetes Mellitus
  * Pre-existing Cardio-vascular Disease including a previous heart attack, stroke, angina or coronary artery bypass surgery of cardiac stents.
  * Pregnancy
  * Smoker
  * Terminal illness
  * Contraindication to gas mask procedure (I.e. Claustrophobia).
  * Chronic Obstructive Pulmonary Disease. (I.e. Chronic Bronchitis or Emphysema).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Blood glucose Area Under the Curve (AUC) | Assessed via 10 blood samples.Two of which will be taken while fasting and the remainder taken at 30, 60, 120 and 180 minutes following both breakfast and lunch meals. This will be assessed for both of the two 7.5 hour experimental treatment conditions.
  Blood glucose AUC refers to the spike of an individuals blood sugar following a meal, the aim of which is to reduce the spike and consequently reduce the area under the curve.

SECONDARY OUTCOMES:
Insulin Area Under the Curve (AUC) | Assessed via 10 blood samples.Two of which will be taken while fasting and the remainder taken at 30, 60, 120 and 180 minutes following both breakfast and lunch meals. This will be assessed for both of the two 7.5 hour experimental treatment conditions.
  Refers to an individuals insulin response to a meal over a prolonged time period during each treatment.
Blood Pressure Area Under the Curve (AUC) | Blood pressure measurements will be taken prior to each blood sample, therefore 10 measurements in total. Two measurements will be taken while fasting and the remainder taken at 30, 60, 120 and 180 minutes following both breakfast and lunch meals.
Cognitive function - Part 1 - Semantic verbal fluency test. | This test will only take one minute in duration. It is administered on arrival at the laboratory (approximately 8am) and will be repeated later on in the day following the last blood sample (approximately 4pm).
  This test assesses semantic memory and language, and participants will be asked to name as many items as they can that belong to a particular category in one minute. For example in the morning, participants will be asked to name as many 'items of clothing', and in the afternoon, they will be asked to name as many 'animals'. This will be done during both experimental conditions so that comparisons can be made.
Cognitive function - Part 2 - Hopkins Verbal Learning test | Participants will undertake this test in the morning, following part 1 of the cognitive test (immediate recall) and also at the end of the experimental day (delayed recall). A maximum of one minute is used to recall as many words as possible.
  This test involves the immediate and delayed recall of a group of 12 words. This is used to assess working memory. Participants will be shown a list of 12 words, from which they must remember and recall as many as possible in the one minute recall period. The participant will have three chances to remember the 12 words in the morning (immediate recall x 3) and then just one chance in the afternoon to recall those remembered during the morning (delayed recall x 1). This will be done during both experimental conditions so that comparisons can be made.
Cognitive function - Part 3 - Trail Making | The time taken to complete this test varies between individuals but on average takes approximately 5 minutes. Participants will undertake this test in the morning, (following part 2 of the cognitive test) and also at the end of the experimental visit.
  Part 3 of the cognitive test assesses cognitive flexibility. For the first part of this test, participants are required to connect randomly located numbers on a screen in numerical order (e.g. 1,2,3,4). For the second part of this test, participants will be expected to connect randomly scattered numbers 'and' letters in numerical 'and' alphabetical order alternately (e.g. 1,A,2,B,3,C). Participants will also be asked to do this as quickly as possible. This will be done during both experimental conditions so that comparisons can be made.
Cognitive function - Part 4 - Rapid Visual Information Processing Test | This part of the test lasts for 5 minutes and will be administered following part 3 of the cognitive test in the morning and also at the end of the experimental day.
  Part 4 of the cognitive test assesses sustained visual attention. This test displays a number on the screen that changes between odd and even digits. Participants must tap the screen each and every time they detect a sequence of three odd or three even consecutive digits. Participants are encouraged to register as many as possible. This will be done during both experimental conditions so that comparisons can be made.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Yates, PhD, Principal Investigator — University of Leicester
Locations (1):
- Leicester Diabetes Centre, Leicester General Hospital, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCarthy M, Edwardson CL, Davies MJ, Henson J, Rowlands A, King JA, Bodicoat DH, Khunti K, Yates T. Breaking up sedentary time with seated upper body activity can regulate metabolic health in obese high-risk adults: A randomized crossover trial. Diabetes Obes Metab. 2017 Dec;19(12):1732-1739. doi: 10.1111/dom.13016. Epub 2017 Jul 20. PMID 28544202